CLINICAL TRIAL: NCT00526994
Title: Randomized Controlled Trial of Routine Screening for Intimate Partner Violence
Brief Title: Randomized Controlled Trial of Routine Screening for IPV
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Joanne Klevens, epidemiologist, Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200-2006-15969/200-2008-28219; IRB #4984; IRB #4985; OMB # 0920-06BM; Contract #200-2008-28219; & 200-2006-15969
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Results first posted 2013-07-31 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Quality of Life; Disability; Utilization of Health Care Services
Keywords: intimate partner violence; domestic violence; spouse abuse; screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Screened (Experimental): Screened w/4 questions on intimate partner violence; if positive, receives referral information
  Interventions: Other: screened
- Universal education (Active Comparator): all participants receive partner violence referral information
  Interventions: Behavioral: universal education
- Control (No Intervention): no screen and no referral

INTERVENTIONS:
Other: screened — Asked 4 questions on current exposure to intimate partner violence; if positive, receives referral information
  Arms: Screened
Behavioral: universal education — receives referral information
  Arms: Universal education

SUMMARY:
This is a randomized controlled trial with three arms to establish the impact of screening and referral to services for women disclosing exposure to IPV.

DETAILED DESCRIPTION:
Approximately 2675 women* will be enrolled and randomized to one of 3 arms. In the first arm, participants will be screened, and if disclosing IPV, will receive information on available resources in the community. In arms two and three, participants will not be screened, but one group will receive information on available resources in the community and the other will not. All three groups will be assessed for quality of life (SF-12;standardized and validated scale with 12 questions that measure overall health (1 item), physical functioning (2 items), role limitations due to physical health problems (4 items), bodily pain (1 item), energy/fatigue (1 item), social functioning (1 item), psychological distress (1 item), and well being (1 item) in the past 4 weeks; items are summed to form a physical health composite scale and a mental health composite scale; each scale is standardized to have a mean of 50 and a standard deviation of 10 for the U.S. population with a possible range from 0 to 100; higher scores represent a better health state); disability; and utilization of health care and IPV services at baseline and at a 12 month follow-up. A pilot study, also using a randomized controlled trial design, will establish the feasibility, acceptability, and impact on disclosure rates, use of referral resources, and potential harms of three screening and referral strategies.

*sample size calculation based n needed to detect a standardized effect size of 0.3 with an α=.05 (1-tailed)and ß=.20 if there's a 20% IPV (+) rate and 30% lost-to-follow-up rate.

ELIGIBILITY:
Inclusion Criteria:

* women attending obstetrics & gynecology (OB-GYN), family planning, general medicine, family medicine or HIV/Sexually transmitted disease (STD) clinic

Exclusion Criteria:

* non-English speaking other than Spanish speakers
* accompanied by a child >3 years of age without adequate provision for child care;
* Visually- or hearing-impaired women;
* without access to a telephone;
* Severe Mental impairment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2700 (Actual)
Dates: Start 2008-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Klevens, MD, PhD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Fantus Health clinic, Chicago, Illinois, United States

REFERENCES:
- [Derived] Klevens J, Sadowski LS, Kee R, Garcia D, Lokey C. Effect of Screening for Partner Violence on Use of Health Services at 3-Year Follow-up of a Randomized Clinical Trial. JAMA. 2015 Aug 4;314(5):515-6. doi: 10.1001/jama.2015.6755. No abstract available. PMID 26241603
- [Derived] Klevens J, Kee R, Trick W, Garcia D, Angulo FR, Jones R, Sadowski LS. Effect of screening for partner violence on women's quality of life: a randomized controlled trial. JAMA. 2012 Aug 15;308(7):681-9. doi: 10.1001/jama.2012.6434. PMID 22893165

RESULTS

PARTICIPANT FLOW:
Recruitment Details: May, 2009-April, 2010 at 10 primary health care clinics in Chicago
Pre-assignment Details: 8 Unenrolled: 7 because computer did not save baseline data & 1 Withdrew
Groups:
- Screened & Referred: Screened w/4 questions on intimate partner violence; if positive, receives referral information
  screening : Asked 4 questions on current exposure to intimate partner violence; if positive, receives referral information
- Universal Education (All Referred): receives referral information
  universal education : receives referral information
Period: Overall Study
Arm/Group | Screened & Referred | Universal Education (All Referred) | Control
Started | 909 | 893 | 898
Completed | 801 | 772 | 791
Not Completed | 108 | 121 | 107
Not completed — Lost to Follow-up | 98 | 108 | 96
Not completed — Death | 4 | 3 | 3
Not completed — Withdrawal by Subject | 2 | 7 | 5
Not completed — incarcerated, impaired, incomplete | 4 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Screened & Referred | Universal Education (All Referred) | Control | Total
Number analyzed (Participants) | 909 | 893 | 898 | 2700
Age Continuous [Mean (Standard Deviation); unit: years] | 39 (15) | 38.3 (14.8) | 38.7 (15.1) | 38.7 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 909 | 893 | 898 | 2700
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life, Physical Health Composite
Description: Assessed with Quality of Life SF-12 V.2 (Ware, Kosinski,Turner-Bowker, & Gandek, 2002). This instrument has 12 items measuring eight subscales of mental and physical health-general health, physical functioning, role limitations due to physical health problems, role limitations due to emotional problems, bodily pain, vitality (energy/fatigue), social functioning, and mental health (psychological distress)-during the past 4 weeks. These subscales are combined to form a physical health composite scale and a mental health composite scale. Each scale is standardized to have a mean of 50 and a standard deviation of 10 for the U.S. population with a possible range from 0 to 100; higher scores represent a better health state.
Time Frame: at one-year follow-up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Screened & Referred | Universal Education (All Referred) | Control
Number analyzed (Participants) | 801 | 772 | 791
units on a scale | 46.8 [46.1 to 47.4] | 46.4 [45.8 to 47.1] | 47.2 [46.5 to 47.8]

2. Secondary Outcome: Utilization of Health Care
Description: number of ambulatory care visits
Time Frame: during past year
Measure: Mean (95% Confidence Interval); unit: visits
Arm/Group | Screened & Referred | Universal Education (All Referred) | Control
Number analyzed (Participants) | 801 | 772 | 791
visits | 5.4 [3.8 to 7.0] | 5.7 [4.1 to 7.3] | 5.9 [4.3 to 7.4]

3. Secondary Outcome: Disability
Description: days lost from housework
Time Frame: one year follow-up
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Screened & Referred | Universal Education (All Referred) | Control
Number analyzed (Participants) | 801 | 772 | 791
days | 1.9 [1.6 to 2.3] | 2.2 [1.8 to 2.5] | 1.9 [1.6 to 2.3]

4. Primary Outcome: Quality of Life, Mental Health Composite
Description: Assessed with the Quality of Life SF-12 v.2 (Ware, Kosinski, Turner-Bowker, & Gandek, 2002). This instrument has 12 items measuring eight subscales of mental and physical health-general health, physical functioning, role limitations due to physical health problems, role limitations due to emotional problems, bodily pain, vitality (energy/fatigue), social functioning, and mental health (psychological distress)-during the past 4 weeks. These subscales are combined to form a physical health composite scale and a mental health composite scale. Each scale is standardized to have a mean of 50 and a standard deviation of 10 for the U.S. population with a possible range from 0 to 100; higher scores represent a better health state.
Time Frame: past 30 days
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Screened & Referred | Universal Education (All Referred) | Control
Number analyzed (Participants) | 801 | 772 | 791
units on a scale | 48.3 [47.5 to 49.1] | 48.0 [47.2 to 48.9] | 47.8 [47.0 to 48.6]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Screened & Referred | Universal Education (All Referred) | Control
Serious Adverse Events (participants affected / at risk) | 0/801 | 0/772 | 0/791
Other Adverse Events (participants affected / at risk) | 0/801 | 0/772 | 0/791

LIMITATIONS AND CAVEATS:
12% lost to follow-up differed in age, education, and insurance status from those retained. Generalizability of the findings is limited by the urban setting; exclusion of some participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes